CLINICAL TRIAL: NCT06085326
Title: Smart Checklist Implementation for Pediatric Tracheal Intubations in the ICU- Multicenter Study
Acronym: SMART PICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 23-021168; R01HS029188 (AHRQ)
Record Dates: First submitted 2023-10-11; First posted 2023-10-16 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Intubation Complication
Keywords: Pediatric; Intubation; PICU; Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Intervention Phase (No Intervention): PICU patients who are intubated without the Smart checklist
- Post-Intervention Phase (Active Comparator): PICU patients who are intubated after implementation of the Smart checklist in the pediatric intensive care unit.
  Interventions: Other: Smart Checklist

INTERVENTIONS:
Other: Smart Checklist — The digitized Smart Checklist includes three new features that currently do not exist on a paper checklist: 1) decision support prompts based on patient-provider dyad characteristics, 2) real time display of patient pertinent airway information from the EHR, and 3) high-risk warning alerts based on predictive analytics with potential explanatory factors from the model.
  Arms: Post-Intervention Phase

SUMMARY:
The purpose of the study is to implement a patient-provider dyad tailored, Electronic Health Record (EHR)-informed, digitized Smart Checklist as a Quality Improvement (QI) intervention to support bedside clinician teams to reduce Adverse Airway Outcomes (AAO) across 6 diverse pediatric intensive care units (ICUs).

DETAILED DESCRIPTION:
More than 20% of the critically ill children who require tracheal intubation suffer from adverse events. To reduce the adverse event risk, and optimize bedside team performance investigators will implement a digitized Smart Checklist that has three specific features: (1) prompts based on patient characteristics, (2) direct display of difficult airway status and airway information, and (3) high-risk warning based on predictive analytics.

This is a stepped-wedge cluster randomized trial of PICU patients who are intubated across 6 participating hospitals to determine if the Smart Checklist reduces the incidence of adverse tracheal intubation associated events.

The primary objective of this study is to determine the clinical impact of the personalized, dynamic, adaptive Smart Checklist implementation on the occurrence of Adverse Airway Outcomes (AAOs) in the pediatric ICU. The secondary objective is to characterize work systems and processes that affect clinical impact of the digitized Smart Checklist.

ELIGIBILITY:
Inclusion Criteria:

All patients intubated in the PICU at participating sites

Exclusion Criteria:

Endotracheal tube exchanges, as this represents a distinct procedure

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Airway Outcomes | During the intubation procedure and up to 20 minutes after procedure
  A composite outcome for adverse events or acute oxygen desaturation <80%

SECONDARY OUTCOMES:
Duration of invasive mechanical ventilation | During the ICU stay, up to 180 days
  Duration of invasive mechanical ventilation (time to extubation or tracheostomy)
Duration of ICU stay | During the ICU stay, up to 180 days
  Duration of ICU stay (days)
ICU mortality | During the ICU stay, up to 180 days
  ICU mortality (all cause)

CONTACTS AND LOCATIONS:
Overall Officials: Akira Nishisaki, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (6):
- United States (6):
  - University of Arkansas, Little Rock, Arkansas
  - Emory University, Atlanta, Georgia
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Akron Children's Hospital, Akron, Ohio
  - Hasbro Children's Hospital, Providence, Rhode Island
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
The PI will share unique research resources developed through this Agency for Healthcare Research and Quality (AHRQ)-funded grant to enhance the value and further the advancement of research. The PI will make data available after study completion and in accordance with AHRQ policies. The data will only be provided to those investigators who agree to adhere to a signed research data use agreement. The execution of the agreement will require approval by the Children's Hospital of Philadelphia (CHOP) Institutional Review Board (IRB) or demonstration of IRB exemption per institutional policy. The data and associated documentation will be available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and does not identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed
Time Frame: Data will be available after study completion
Access Criteria: The data and associated documentation will be available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and does not identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed